CLINICAL TRIAL: NCT05799859
Title: Treatment of Local Gingival Recession With an Enamel Matrix Protein Coated Collagen Matrix - a Randomized Controlled Trial
Brief Title: Treatment of Local Gingival Recession With an Enamel Matrix Protein Coated Collagen Matrix
Acronym: EmdoDerm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EmdoDerm
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Gingival Recession
Keywords: coronally advanced flap; collagen; enamel matrix protein; dental enamel protein; gingival recession; periodontal plastic surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF + CM (Active Comparator): Coronally advanced flap (CAF) and collagen matrix (CM)
  Interventions: Device: Use of coronally advanced flap (CAF) and collagen matrix (CM)
- CAF + CM +EMD (Experimental): Coronally advanced flap (CAF), collagen matrix (CM) and additional application of enamel matrix derivatives (EMD).
  Interventions: Device: Use of coronally advanced flap (CAF) and collagen matrix (CM) and additional application of enamel matrix derivatives (EMD).

INTERVENTIONS:
Device: Use of coronally advanced flap (CAF) and collagen matrix (CM)
  Arms: CAF + CM
Device: Use of coronally advanced flap (CAF) and collagen matrix (CM) and additional application of enamel matrix derivatives (EMD).
  Arms: CAF + CM +EMD

SUMMARY:
The clinical trial studies patients with gingival recession defects (receding gums).

The goal of the study is to test whether the additional use of enamel matrix derivatives (EMD), combined with the use of a coronally advance flap (CAF) and a CM (collagen matrix), shows a better outcome compared to a comparison group. The comparison group comprises patients receiving treatment with CAF and CM without the use of EMD.

DETAILED DESCRIPTION:
The study aims to evaluate the influence of the additional use of EMD in treatment of gingival recession defects using a coronally advance flap (CAF) and a CM (collagen matrix) by means of digital and clinical assessment methods. The reference group comprises patients receiving treatment with CAF and CM without the application of EMD.

In this prospective, randomized, controlled study, recession height and area, width and thickness of keratinized gingiva, pocket probing depth, and the clinical attachment level were measured at baseline and followed-up for one year.

15 patients with 24 gingival recession defects (Recession Type 1 after Cairo/Miller Class I or II) were recruited and were randomly assigned into the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* able to achieve good oral hygiene (full mouth plaque score < 20 %, full mouth bleeding score < 20%),
* patients presenting with at least one gingival recession defect

Exclusion Criteria:

* general contraindications to dental surgery under local anaesthesia (e.g., severe systemic diseases, tumours, severe cardiovascular diseases, uncontrolled diabetes mellitus);
* ongoing or previous chemotherapy, radiotherapy, or bisphosphonate therapy;
* self-reported heavy smokers (more than 10 cigarettes/day);
* pregnancy and nursing mothers;
* disorders or treatments that impair wound healing;
* long-term treatment with high-dose steroids or anticoagulants;
* bone metabolism disorders;
* infections or vascular disorders in the region to be treated;
* known hypersensitivity to porcine collagen;
* patients with severe peripheral artery disease or autoimmune diseases;
* extruded or malpositioned teeth.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Gingival recession height | 12 months postoperatively
  Gingival recession height in millimeters, measured as the distance from cementoenamel junction to gingival margin

SECONDARY OUTCOMES:
Width of keratinized tissue (WKT) | 12 months postoperatively
  Width of keratinized tissue in millimeters, .as distance between gingival margin and muco-gingival junction
pocket probing depth (PPD) | 12 months postoperatively
  Pocket probing depth in millimeters, measured as the distance from gingival margin to bottom of gingival sulcus
Clinical attachment loss (CAL) | 12 months postoperatively
  Clinical attachment loss in millimeters

IPD SHARING:
Plan to Share IPD: No